CLINICAL TRIAL: NCT03945500
Title: Assessment of a Standardized Home Spirometry Method for Frequent Monitoring of Lung Function in a Normal Population
Brief Title: Standardized Home Spirometry Method in Normal Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 201806011
Record Dates: First submitted 2019-05-01; First posted 2019-05-10 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Mobile Applications; Healthy Volunteers; Feasibility Study

STUDY DESIGN:
Intervention Model Description: Evaluate the feasibility of using a Standardized Home Spirometry Method and associated investigational Home Spirometry Mobile Medical Software (IT App) and Server "Dashboard" in a healthy volunteer population before beginning a separate full clinical trial in the lung transplant population. Feasibility of using the Standardized Home Spirometry Method and associated Home Spirometry Mobile Medical Software (IT App and Server "Dashboard" to develop normal range values, to detect a value outside of the normal range, to evaluate a value outside of the normal range with a symptom survey and to download all data to a Central Monitoring Institute will be evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standardized Home Spirometry (SHS) Method (Experimental): The Standardized Home Spirometry (SHS) Method consists of an Investigational Mobile Medical Application embedded in an Android Tablet & FDA approved spirometer & pulse oximeter.
  Participants will be trained with the SHS method, perform an initial home spirometry test session & a lab-based spirometry test (if practicable).
  Pre-surveillance Phase:Daily SHS Testing for 4 to 10 weeks to enable the Mobile Medical application to generate volunteer specific normal range.
  Surveillance Phase: At least weekly SHS Testing. During approximately two months of the surveillance phase, the volunteer will test one to four times per week to assess the SHS neural pathways as directed by the study team. Test sessions will be documented on a test log. Subjects may be asked to perform additional SHS pathway test logs, continue at least weekly testing, pause testing or end participation following completion of the initial SHS neural pathway test log.
  Interventions: Device: Investigational Mobile Medical Software Application & IT Dashboard Application, FDA approved Bluetooth spirometer, FDA approved pulse oximeter

INTERVENTIONS:
Device: Investigational Mobile Medical Software Application & IT Dashboard Application, FDA approved Bluetooth spirometer, FDA approved pulse oximeter — Standardized Home Spirometry (SHS) Method consists of an Investigational Mobile Medical Application embedded into an Android Tablet, an FDA approved Bluetooth spirometer, an FDA approved pulse oximeter. HIPAA compliant data will be sent to an Investigational IT dashboard maintained at the Central Monitoring Institute Server.
  Volunteers will train in-center or remotely & perform baseline testing with the SHS method along with a baseline laboratory-based spirometry test (if practicable).
  Pre-Surveillance Phase: Daily home spirometry method testing for 4 to 10 weeks to enable normal range calibration.
  Surveillance Phase: At least weekly home spirometry method testing for 2-10 months of participation. Volunteers will maintain a test log during study team directed SHS software pathway functionality testing.
  Other Names: Baseline Laboratory Spirometry Testing

SUMMARY:
This study was designed to evaluate the feasibility of using a Standardized Home Spirometry (SHS) Method to develop normal range values, to detect a variance (i.e., a value outside of that normal range), to evaluate a variance with a questionnaire, and to download all data in normal volunteers prior to evaluation and use on a larger scale for lung transplant recipients. The Standardized Home Spirometry (SHS) Method consists of a FDA-approved Bluetooth Spirometry unit, FDA approved Bluetooth Pulse Oximeter and an Android-based Tablet which is embedded with an investigational Home Spirometry Mobile Medical Software Application for data and symptom survey collection and transmission over secure WiFi or cellular connectivity in HIPAA compliant fashion (labeled only with a date/time and machine ID stamp) to an associated investigational IT Server Dashboard at the Central Monitoring Institute Server at Washington University in St. Louis.

DETAILED DESCRIPTION:
Study Objective: This study was designed to evaluate the feasibility of use of a Standardized Home Spirometry(SHS) Method using a Home Spirometry Monitoring Kit consisting of FDA-approved Blue-tooth Spirometry unit, Blue-tooth pulse oximeter and an Android-based Tablet with an embedded investigational home spirometry mobile medical software application for data and symptom survey collection and transmission over secure WiFi or cellular data transmission portal in HIPAA compliant fashion to an associated investigational IT dashboard application at the Central Monitoring Institute (CMI) Server at Washington University in St. Louis, to develop normal range values, to detect a variance (i.e., a value outside of that normal range), to evaluate a variance with a questionnaire, and to download all data to the CMI in a small pilot of healthy volunteers prior to evaluation and use on a larger scale for lung transplant recipients.

The investigational IT application will monitor lung function but do nothing more than collect data. It will adjust monitoring frequency and trigger physician review of home spirometry results at a more frequent interval but will not be directly involved in decisions regarding diagnosis or treatment.

Study Type: Non-randomized, single-arm, prospective cohort study

Intervention:

* The Home Spirometry Monitoring System will consist of:

  * FDA approved Blue tooth Spirometry unit
  * FDA approved pulse oximeter
  * An Android-based tablet with embedded investigational mobile medical software application for symptom survey/data collection and data processing and transmission
* WiFi or cellular connectivity to be used for data transmission and communication between an Android Pad and an associated Investigational server dashboard application at the Central Monitoring Institute
* Normal Volunteer Monitoring Data is sent in a HIPAA compliant fashion (data with date/time stamp and device ID only) to a Central Monitoring Institute (CMI) server maintained at Washington University in St. Louis
* Participants will undergo training to activate and use the Home Spirometry Monitoring System.
* Data evaluation by a pulmonologist within CMI:

  * Trend analysis on a monthly basis and
  * When a variance is detected with or without potentially associated symptoms.
  * A monthly summary report
* Participants may undergo one Laboratory-based Spirometry Test (if practicable) and perform a test session using the standardized home spirometry method system at baseline.
* Participation may last up to one year.

Standardized Home Spirometry testing interval at least weekly with an initial testing period of greater frequency to enable normal range calibration. Volunteers will require initial in center or remote training with the Standardized home spirometry method & performance of baseline home spirometry method testing and a (baseline) laboratory-based spirometry test (if practicable).

Pre-Surveillance Phase: Daily home spirometry method measurements for 4 to 10 weeks to enable normal range calibration. Volunteers who have either a statistically significant (p-value <0.01) rate of change in FEV1 or a change in FEV1 rate of decline that exceeds an absolute value (+/-) of 30 mL/month using home spirometry based FEV1 values obtained during the normal range development period are not eligible to advance to the Surveillance Phase and may be discontinued from the study.

Surveillance Phase: At least weekly home spirometry method measurements for two to ten months of participation. An FEV-1 (Forced Expiratory Volume in one second) variance is defined as an FEV-1 value that is outside the 95% CI (Confidence Interval) of the participant's normal FEV-1 reference range that was determined immediately after enrollment.

If an FEV-1 variance is detected by the Android Pad, the IT application automatically requests that the participant complete a symptom survey. This information when used in combination with other data will result in initiation of the following actions:

If an FEV-1 variance is categorized as being suspicious for acute medical illness by the CMI (i.e., with clinical symptoms consistent with upper or lower respiratory infection/CHF), the spirometry data and participant survey responses will trigger overview by the CMI laboratory staff and if deemed suspicious for acute medical illness results will be made accessible to the participant's designated health professionals. If critical values or clinical symptoms are obtained consistent with urgent compromise (e.g., evidence of hypoxemia or respiratory distress), the CMI (PFT (Pulmonary Function Testing) Laboratory staff pulmonologist) will make timely attempts to reach the participant or participant's health professionals. In this study, this is expected to be an exceedingly rare occurrence, and most likely would not occur at all. If acute medical illness has been ruled in, participant spirometry surveillance will be reinitiated after an appropriate period of treatment, which will be determined by the participant's managing physician who will notify CMI when the participant has recovered from their acute illness.

Variance not suspicious for acute medical illness with no apparent clinical symptoms consistent with infection/CHF: if supplemental questionnaire or clinical data is not consistent with an acute medical illness, the following actions will be taken:

Persistence Evaluation: Participants will be directed to obtain daily spirometric measurements along with repeated completion of the questionnaire for a total of 4 consecutive days CMI Pulmonology Review: Consistently low Spirometry values (persistence) will prompt early review of these values along with previous Spirometry history by CMI pulmonology staff.

Random Symptom Surveys may also generate (in the absence of a variance) however only Symptom Surveys prompted by Variances will result in further action as described above.

During the first two months (approximately) of Surveillance, Volunteers will be directed to intentionally induce variances, symptoms, incomplete connections/testing/survey, etc., in order to fully test and assess the functionality of the Mobile Medical Software neural pathways (IT app and Dashboard server) as directed by the study team. Volunteers will document test on a test log.

The FDA issued a non-significant risk (NSR) device study letter on 12/3/2018 for the Home Spirometry Mobile Medical Software.

ELIGIBILITY:
Inclusion Criteria:

1. Age (18 years old or older)
2. Volunteers who provide written informed consent to participate in this study and who are willing and able to perform frequent home spirometry monitoring and laboratory-based spirometry if practicable, per protocol.

Exclusion Criteria:

1. Known cardiac, pulmonary or other condition, that may interfere with the subject's ability to perform lab-based pulmonary function testing or standardized home spirometry.
2. Any condition that would significantly affect the participant's ability to adhere to the protocol, or affect interpretation of the study results.
3. Pregnant or planning to become pregnant during the study. Pregnant volunteers are excluded as changes in spirometry associated with a gravid uterus could alter outcome data. (Volunteers should take measures to prevent pregnancy while participating in the study.)
4. Inability to provide informed consent or to comply with study assessments (e.g. due to cognitive impairment or geographic distance, lack of WiFi and/or cellular access or inadequate English literacy/comprehension to operate the Home Spirometry System)
5. Concomitant participation in another trial with an investigational device or investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of using the Standardized Home Spirometry (SHS) Method and associated IT Dashboard Server: Assess Home Spirometry reproducibility during pre-surveillance period. | Up to 8 weeks
  Evaluate daily FEV1 variability between replicate measurements by summarizing between measurement %difference; Evaluate between day variability in highest FEV1 (FEV1 Max) variability by summarizing %Difference from FEV1 Max values and two SD (Standard Deviation) Coefficient of Variation (expected to be less than 30%) between FEV1 measurements during pre-surveillance period.
Feasibility of using the Standardized Home Spirometry (SHS) Method and associated IT Dashboard Server: Drift Assessment | Up to 8 weeks
  Evaluate the functionality of the investigational Mobile Medical Software Application and associated IT Server Dashboard for statistically significant drift in relationship between %FEV1 Max or mean FEV1 Max over time and subsequent transition to Surveillance monitoring stage.
Feasibility of using the Standardized Home Spirometry (SHS) Method and associated IT Dashboard Server: Pathway Verification | Through study completion, up to 10 months
  Evaluate the Mobile medical application software and associated IT server data processing pathways using % initial error rate (initial error rate and subsequent error rate, after any potential adjustments are made in mobile medical application if changes are required).

CONTACTS AND LOCATIONS:
Overall Officials: George Despotis, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yusen RD, Edwards LB, Kucheryavaya AY, Benden C, Dipchand AI, Dobbels F, Goldfarb SB, Levvey BJ, Lund LH, Meiser B, Stehlik J; International Society for Heart and Lung Transplantation. The registry of the International Society for Heart and Lung Transplantation: thirty-first adult lung and heart-lung transplant report--2014; focus theme: retransplantation. J Heart Lung Transplant. 2014 Oct;33(10):1009-24. doi: 10.1016/j.healun.2014.08.004. Epub 2014 Aug 14. No abstract available. PMID 25242125
- [Background] Meyer KC, Raghu G, Verleden GM, Corris PA, Aurora P, Wilson KC, Brozek J, Glanville AR; ISHLT/ATS/ERS BOS Task Force Committee; ISHLT/ATS/ERS BOS Task Force Committee. An international ISHLT/ATS/ERS clinical practice guideline: diagnosis and management of bronchiolitis obliterans syndrome. Eur Respir J. 2014 Dec;44(6):1479-503. doi: 10.1183/09031936.00107514. Epub 2014 Oct 30. PMID 25359357
- [Background] Kapila A, Baz MA, Valentine VG, Bhorade SM; AIRSAC investigators. Reliability of diagnostic criteria for bronchiolitis obliterans syndrome after lung transplantation: a survey. J Heart Lung Transplant. 2015 Jan;34(1):65-74. doi: 10.1016/j.healun.2014.09.029. Epub 2014 Oct 7. PMID 25447585
- [Background] Slovis BS, Loyd JE, King LE Jr. Photopheresis for chronic rejection of lung allografts. N Engl J Med. 1995 Apr 6;332(14):962. doi: 10.1056/NEJM199504063321417. No abstract available. PMID 7877665
- [Background] O'Hagan AR, Stillwell PC, Arroliga A, Koo A. Photopheresis in the treatment of refractory bronchiolitis obliterans complicating lung transplantation. Chest. 1999 May;115(5):1459-62. doi: 10.1378/chest.115.5.1459. PMID 10334173
- [Background] Salerno CT, Park SJ, Kreykes NS, Kulick DM, Savik K, Hertz MI, Bolman RM 3rd. Adjuvant treatment of refractory lung transplant rejection with extracorporeal photopheresis. J Thorac Cardiovasc Surg. 1999 Jun;117(6):1063-9. doi: 10.1016/s0022-5223(99)70241-2. PMID 10343253
- [Background] Villanueva J, Bhorade SM, Robinson JA, Husain AN, Garrity ER Jr. Extracorporeal photopheresis for the treatment of lung allograft rejection. Ann Transplant. 2000;5(3):44-7. PMID 11233043
- [Background] Benden C, Speich R, Hofbauer GF, Irani S, Eich-Wanger C, Russi EW, Weder W, Boehler A. Extracorporeal photopheresis after lung transplantation: a 10-year single-center experience. Transplantation. 2008 Dec 15;86(11):1625-7. doi: 10.1097/TP.0b013e31818bc024. PMID 19077900
- [Background] Morrell MR, Despotis GJ, Lublin DM, Patterson GA, Trulock EP, Hachem RR. The efficacy of photopheresis for bronchiolitis obliterans syndrome after lung transplantation. J Heart Lung Transplant. 2010 Apr;29(4):424-31. doi: 10.1016/j.healun.2009.08.029. Epub 2009 Oct 22. PMID 19853479
- [Background] Jaksch P, Scheed A, Keplinger M, Ernst MB, Dani T, Just U, Nahavandi H, Klepetko W, Knobler R. A prospective interventional study on the use of extracorporeal photopheresis in patients with bronchiolitis obliterans syndrome after lung transplantation. J Heart Lung Transplant. 2012 Sep;31(9):950-7. doi: 10.1016/j.healun.2012.05.002. PMID 22884382
- [Background] Greer M, Dierich M, De Wall C, Suhling H, Rademacher J, Welte T, Haverich A, Warnecke G, Ivanyi P, Buchholz S, Gottlieb J, Fuehner T. Phenotyping established chronic lung allograft dysfunction predicts extracorporeal photopheresis response in lung transplant patients. Am J Transplant. 2013 Apr;13(4):911-918. doi: 10.1111/ajt.12155. Epub 2013 Feb 13. PMID 23406373
- [Background] Del Fante C, Scudeller L, Oggionni T, Viarengo G, Cemmi F, Morosini M, Cascina A, Meloni F, Perotti C. Long-Term Off-Line Extracorporeal Photochemotherapy in Patients with Chronic Lung Allograft Rejection Not Responsive to Conventional Treatment: A 10-Year Single-Centre Analysis. Respiration. 2015;90(2):118-28. doi: 10.1159/000431382. Epub 2015 Jun 20. PMID 26112178
- [Background] Liistro G, Vanwelde C, Vincken W, Vandevoorde J, Verleden G, Buffels J; COPD Advisory Board. Technical and functional assessment of 10 office spirometers: A multicenter comparative study. Chest. 2006 Sep;130(3):657-65. doi: 10.1378/chest.130.3.657. PMID 16963659
- [Background] Lefebvre Q, Vandergoten T, Derom E, Marchandise E, Liistro G. Testing spirometers: are the standard curves of the american thoracic society sufficient? Respir Care. 2014 Dec;59(12):1895-904. doi: 10.4187/respcare.02918. Epub 2014 Sep 2. PMID 25185146